CLINICAL TRIAL: NCT06649474
Title: Evaluation, in Humans, of the Correlation Between Hepatotoxicity, Neurotoxicity Induced by Oxaliplatin, and Blood Levels of HMGB1
Acronym: HEPATOXALI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2023 JARY; 2023-A02427-38 (Other: registration number with the French drug agency)
Record Dates: First submitted 2024-09-05; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer; Resectable Pancreatic Adenocarcinoma; Adenocarcinoma; Resectable Esophageal Cancer; Resectable Gastric or Gastroesophageal Junction Adenocarcinoma; Oesophagogastric Cancer
Keywords: resecable pancreatic, oesophageal, gastric or gastroesophageal junction adenocarcinoma.; Patients able to have a laparoscopy; chemotherapy before surgery
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: 50 patients with pancreatic adenocarcinoma and 50 patients with oesogastric adenocarcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- comparate the Serum HMGB1 concentrations between patients with grade <2 SOS and those with grade 2,3 (Other)
  Interventions: Biological: assess the serum HMGB1 concentrations before and after an oxaliplatin-based chemotherapy

INTERVENTIONS:
Biological: assess the serum HMGB1 concentrations before and after an oxaliplatin-based chemotherapy — assess the serum HMGB1 concentrations

SUMMARY:
Oesogastric and pancreatic adenocarcinomas are poor-prognosis cancers. Incidence of pancreatic cancer drastically increases to such an extent that it will become the second cause of cancer's mortality by 2030. A major challenge is to optimize the therapies for localized setting, when oxaliplatin-based chemotherapy is the standard, before and after surgical excision. Because in 50% of cases oxaliplatin triggers a grade 2-3 sinusoidal obstruction syndrome (SOS) which increases post-operative morbidity, decreases histological response to chemotherapy, increases tumor recurrence, and aggravates the risk of chemotherapy-induced peripheral neuropathy (CIPN).

There is an urgent need to better understand the biological processes involved in SOS, in order to prevent and treat it without stopping or reducing oxaliplatin administration.

The biological link between oxaliplatin and SOS has not been described, but recent murine experiments argue for HMGB1 to be the mediator released after exposure to oxaliplatin and inducing SOS, and thereafter CIPN. To date, no biomarker is established between murine and patient analyses, and the release of HMGB1 after oxaliplatin treatment and its effect on hepatic parenchyma is not described in patients. Investigators hypothesized is that HMGB1 would also been increased in patients after oxaliplatin treatment, and correlated to the development of SOS and CIPN. If confirmed, personalized treatment will be possible to target this pathway.

Therefore, investigators propose to dynamically explore this hypothesis in localized oesogastric and pancreatic cancer patients who will be routinely managed by an initial laparoscopy and post-oxaliplatin surgical excision.

ELIGIBILITY:
Inclusion Criteria:

* ECOG WHO Performance status = 0 or 1
* Signed and dated informed consent
* Patients with histological diagnosis of oesogastric or pancreatic adenocarcinoma
* Resectable tumors
* Patients able to have a laparoscopy
* In case of absence of peritoneal invasion on the laparoscopy, patient candidate to a chemotherapy schedule by FLOT or FOLFOX in perioperative setting for oesogastric adenocarcinoma, or FOLFIRINOX in perioperative setting for pancreatic adenocarcinoma
* Registration in a national health care system (CMU included)
* Patient speak and understand the french

Exclusion Criteria:

* Histology other than adenocarcinoma
* Metastatic disease
* History of previous treatment with oxaliplatine
* History of systemic chemotherapy administration within 5 years prior to inclusion,
* Patient with an non balanced progressive condition/disease (liver failure, renal failure (creatinine clearance <30mL/min), respiratory failure, congestive heart failure, myocardial infarction in the last 6 months, etc.),
* Patient on curative dose anticoagulant,
* Patient with complete dihydropyrimidine dehydrogenase deficiency (Uracilemia ≥ 150 ng/ml),
* Patient not operable for the pathology concerned,
* Pregnant or breastfeeding woman, woman of childbearing age who has not performed a pregnancy test before the procedure,
* Patient with legal incapacity (person deprived of liberty or under curatorship, stutorship, safeguard of justice),
* Patient who, for psychiatric, social, family or geographical reasons, cannot be followed and/or comply with the requirements of the study,,
* Discovery of peritoneal invasion during the peritoneal exploratory of the laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum HMGB1 concentrations | At exploratory laparoscopy and at the surgery
  Assess Serum HMGB1 concentrations in two groups of patients : with grade 0 or 1 SOS and with grade ≥2 SOS, at two timepoints: before exploratory laparoscopy and before surgical excision to determinate the effect of HMGB1 on SOS development

SECONDARY OUTCOMES:
variation of serum HMGBI concentration (ng/ml) | at the exploratory laparoscopy, at the first (Day1) and last cycle (assessed up to 75 days) of chemotherapy before surgery (each cycle=14 days) and at the surgery
  mesurated the serum HMGB1 concentration (ng/ml) at several time of treatment of the patient then comparated these assess the dynamic variation of serum HMGB1 concentrations after oxaliplatin-based chemotherapy in oesogastric and pancreatic cancer patients with grade 0 or 1 SOS and with grade ≥2 SOS
variation of serum RAGE (receptor of HMGBI) concentration | at the exploratory laparoscopy, at the first (Day1) and last cycle (assessed up to 75 days) of chemotherapy before surgery (each cycle=14 days) and at the surgery
  mesurated the serum RAGE concentration (ng/ml) at several time of treatment of the patient then comparated these assess the dynamic variation of serum HMGB1 concentrations after oxaliplatin-based chemotherapy in oesogastric and pancreatic cancer patients with grade 0 or 1 SOS and with grade ≥2 SOS
sinusoidal obstruction syndrome (SOS) diagnosis | before to began chemotherapy and from 15 to 21 days after the last cycle of chemotherapy before surgery
  compare SOS histology diagnosis (absent, mild, moderate, severe) with no invasive biological scores "APRI and FIB4"which use ASAT (U/L), ALAT(U/L), plaquettes (G/L) and the age (years) of the patient
sinusoidal obstruction syndrome (SOS) diagnosis | before to began chemotherapy and from 15 to 21 days after the last cycle of chemotherapy before surgery
  compare SOS histology diagnosis (absent, mild, moderate, severe)) with splenic's volumetric measured by radiological's assessment
Evaluated the chemotherapy-induced peripheral neuropathy (CIPN) | at the first (Day1) and last cycle (assessed up to 75 days) of chemotherapy before surgery (each cycle=14 days); at the surgery and at the first cycle (D1) then last cycle (assessed up to 75 days) after surgery
  the CIPN will be evaluate by the investigator who used the CTCAEv5 classification.
Evaluated the chemotherapy-induced peripheral neuropathy (CIPN) | at the first (Day1) and last cycle (assessed up to 75 days) of chemotherapy before surgery (each cycle=14 days); at the surgery and at the first cycle (D1) then last cycle (assessed up to 75 days) after surgery
  the CIPN will be evaluate by each patient who completed the CIPN20 questionnary
Evaluated the chemotherapy-induced peripheral neuropathy (CIPN) | at the first (Day1) and last cycle (assessed up to 75 days) of chemotherapy before surgery (each cycle=14 days); at the surgery and at the first cycle (D1) then last cycle (assessed up to 75 days) after surgery
  the CIPN will be evaluate by each patient who completed the visual analog score for pain
Predictive value of HMGB1 for the development of SOS and CIPN | from exploratory laparoscopy to last cycle of chemotherapy after surgery assessed up to 10 month
  Correlate CIPN, neuropathic pain with SOS, HMGB1, and RAGE measurements

CONTACTS AND LOCATIONS:
Overall Officials: Marine JARY, MD, Principal Investigator — CHU Estaing de Clermont Ferrand/FRANCE
Locations (1):
- CHU Estaing de Clermont-Ferrand, Clermont-Ferrand, France